CLINICAL TRIAL: NCT07258043
Title: Efficacy on Progression Free Overall Survival of a Dose-Adjusted Regimen in Frail Adult Patients With Acute Lymphoblastic Leukemia
Brief Title: Efficacy of Dose-Adjusted Regimen on Survival in Frail Adults With Acute Lymphoblastic Leukemia
Acronym: EPOCH
Status: Recruiting | Type: Observational
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Christian Omar Ramos-Peñafiel, MD, PhD, Medical Doctor, Principal Investigator, Clinical Professor, Hospital General de México Dr. Eduardo Liceaga
Other Study IDs: HGMexicoEduardoLiceaga
Record Dates: First submitted 2025-08-27; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Acute Lymphobkastic Leukemia; Leukemia; Overall Survival
Keywords: acute lymphoblastic leukemia; EPOCH
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Palliative Care; Blood Transfusion; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Bone marrow biopsy will be retained
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Frail ALL patients by ECOG >1 or KPS <80%, or with severe toxicity from induction therapy: Patients newly diagnosed with acute lymphoblastic leukemia (ALL) who are considered clinically frail based on an ECOG performance status score greater than 1 or a Karnofsky score below 80%, indicating a high risk of severe chemotherapy-related toxicity. This group also includes patients who have previously received induction therapy and experienced severe, limiting toxicity that prevents continuation of intensive treatment regimens. These criteria identify a vulnerable population for whom standard chemotherapy may not be suitable, necessitating alternative, less intensive treatment approaches to reduce toxicity while maintaining therapeutic efficacy
  Interventions: Drug: Patients meeting criteria will receive DA-EPOCH via central line for 5 days every 21 days, with monitoring, supportive care, transfusions, prophylaxis, and G-CSF for 5 doses per cycle

INTERVENTIONS:
Drug: Patients meeting criteria will receive DA-EPOCH via central line for 5 days every 21 days, with monitoring, supportive care, transfusions, prophylaxis, and G-CSF for 5 doses per cycle — After patient selection and confirmation of inclusion criteria, the DA-EPOCH treatment regimen will be initiated. It is typically administered through a central line over 5 days, during which adverse events will be closely monitored. Each treatment cycle lasts 21 days. All patients will receive the same level of care as those undergoing high-intensity chemotherapy, including monitoring of transfusion needs, supportive care with prophylactic medications, and the administration of colony-stimulating factors, with a total of 5 doses per cycle. The treatment regimen consists of six cycles, during which intrathecal chemotherapy will be administered to prevent central nervous system relapse. This prophylaxis will be given between each cycle. After completing the six cycles, patients will continue with a maintenance regimen consisting of 6-mercaptopurine at 50 mg/m² of body surface area from Monday to Friday, along with weekly intramuscular methotrexate (50 mg), total duration for 2 years

SUMMARY:
Acute lymphoblastic leukemia (ALL) is characterized by the abnormal proliferation of immature precursor cells, disrupting normal hematopoiesis and causing severe anemia and thrombocytopenia due to genetic mutations. Conventional treatment with intensive chemotherapy is limited for elderly patients or those with comorbidities, adversely affecting their survival. In Mexico, alongside a higher incidence, treatment-related complications are more frequent, particularly with drugs such as asparaginase or anthracyclines, which limits therapeutic efficacy. The transition to infusion-based therapies promises to reduce these complications, improve treatment tolerance, and optimize clinical outcomes, marking a significant advancement in the management of this disease. Modifying treatment regimens toward infusion therapies has the potential to significantly reduce adverse complications, enhance treatment tolerance, and ultimately improve clinical outcomes for patients who cannot benefit from conventional intensive regimens. This approach not only aims to optimize treatment effectiveness but also to minimize associated risks, thus representing an important advancement in the management of acute lymphoblastic leukemia in clinical settings such as those in Mexico

DETAILED DESCRIPTION:
The treatment of acute lymphoblastic leukemia (ALL) in adults represents a therapeutic challenge, particularly in patients with high-risk factors, clinical frailty, or socioeconomic limitations that hinder adherence to intensive outpatient regimens. While protocols such as HyperCVAD have been widely used, their toxicity can be significant in certain subgroups. In this context, the EPOCH regimen has been explored as an inpatient consolidation alternative that allows a gradual transition toward less toxic regimens, with potential benefits in vulnerable populations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute lymphoblastic leukemia (ALL) according to the World Health Organization (WHO) criteria
* Older than 18 years old
* ECOG Performance Status Scale >1 or the Karnofsky Performance Status (KPS) <80%.
* Comorbidities: diabetes mellitus, arterial hypertension, thrombotic events, endocrine disorders, or any condition that hinders the administration of full-dose chemotherapy.
* Toxicity prior to a standard chemotherapy regimen.
* Both genders
* Over 18 years of age
* No upper age limit
* Signed informed consent

Exclusion Criteria:

´- Patients refractory to induction treatment

* Patients who have previously received a low-intensity regimen due to comorbidities
* Biphenotypic leukemia
* CNS involvement at diagnosis requiring radiotherapy
* Patients whose survival is expected to be less than 48 hours due to leukemiarelated complications
* Patients with a history of ischemic or hemorrhagic stroke or severe neurological deterioration
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a de novo diagnosis of acute lymphoblastic leukemia, considered frail according to the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale or with a Karnofsky Performance Score below 80%, indicating a high risk of severe chemotherapy-related toxicity, or patients who have received induction therapy and experienced severe and limiting toxicity.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-07-23 (Estimated); Study Completion 2026-07-26 (Estimated)

PRIMARY OUTCOMES:
To determine the proportion of overall survival and disease-free survival | From enrollment until 1 year after the end of treatment.
  For the survival analysis, the Kaplan-Meier method will be used, which is a non-parametric technique employed to estimate the survival function from time-to-event data.

SECONDARY OUTCOMES:
To determine the proportion of complete remissions (<5% blasts per field) after the first 4 weeks of induction therapy and the proportion of measurable residual disease (proportion of cells) at 6 weeks. | Complete Remision (CR) at 4 weeks after induction and measurable residual disease (MRD) at 6 weeks of treatment.
  Complete remission (CR) will be evaluated by bone marrow aspiration and optical microscopy review at 4 weeks after induction, while measurable residual disease (MRD) will be assessed also by bone marrow aspiration ans measured by flow cytometry at 6 weeks of treatment.
To establish the proportion of serious adverse events associated with the chemotherapy regimen. | From enrollment until 1 year after the end of treatment.
  These will be graded according to the adverse events scale. The National Comprehensive Cancer Network (NCCN) adverse events scale, known as the 'NCCN Common Terminology Criteria for Adverse Events' (NCCN CTCAE), is a tool used to classify the severity of adverse events that occur during clinical trials of cancer treatments.
To describe the proportion of severe neutropenia events and treatment-related mortality | From enrollment until 1 year after the end of treatment.
  Neutropenia events associated with chemotherapy will be quantified in each cycle, and their proportion will be established per administered cycle
To describe the length of hospital stay in days. | From hospital admission to the last day of stay for each administered cycle (each cycle is 21 days).
  The days of hospital stay will be quantified for each cycle of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Christian O Ramos, MD, Principal Investigator — Hospital General de México Dr. Eduardo Liceaga
Locations (1):
- Hospital General de México Dr. Eduardo Liceaga, Mexico City, Mexico City, Mexico